CLINICAL TRIAL: NCT05594173
Title: Chewing and Oral Processing of Solid Food in Healthy Swallowing
Brief Title: Chewing and Oral Processing of Solid Food
Acronym: NIH_HVX6
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-9431.10; R01DC011020 (NIH)
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Food texture modification — Food prepared in three different consistencies: minced and moist, soft and bite-sized and regular, as defined by the International Dysphagia Diet Standardisation Initiative

SUMMARY:
Food texture modification is commonly used as an intervention for people with dysphagia (swallowing impairment). However, the field currently lacks a proper understanding of how this intervention works. The overall goal of this project was to collect measurements of food bolus transit through the oropharynx (i.e., mouth and throat) during chewing, oral processing and swallowing.

DETAILED DESCRIPTION:
Aim: To explore chewing and oral processing behaviors across solid foods of different consistencies (minced and moist, soft & bite-sized, regular).

Healthy adult participants will be asked to swallow foods representative of the "minced and moist", "soft and bite-sized" and "regular" consistency levels of the International Dysphagia Diet Standardisation Initiative.

We will measure the number of chews taken per bolus and the overall duration of chewing to understand differences across consistencies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults under age 60

Exclusion Criteria:

* prior history of swallowing, motor speech, gastro-esophageal or neurological difficulties, chronic sinusitis or taste disturbance.
* history of surgery to the speech or swallowing apparatus (other than routine tonsillectomy or adenoidectomy)
* Type 1 Diabetes
* Current use of dentures
* cognitive communication difficulties that may hinder comprehension of the study documents or instructions
* known allergies to medical adhesive
* known allergies to ingredients of the food products used in the experiment .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers with no history of swallowing difficulty
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona M Steele, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants: Healthy adults with no history of difficulties with chewing or swallowing.
Period: Overall Study
Arm/Group | Healthy Participants
Started | 20
Completed | 17
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — COVID-19 Pandemic | 2

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Participants
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 26 [22 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Chewing Cycles Per Bolus
Description: Using surface electromyography (sEMG) of the masseter muscle, we will count the number of muscle contraction spikes (i.e. chewing cycles) seen for chewing activity for a single comfortable bite of each bolus type.
Time Frame: Baseline (single timepoint only)
Population: Data for 3 additional participants could not be analyzed due to poor electromyography signal quality.
Measure: Mean (Standard Deviation); unit: number of chewing cycles
Groups:
- Healthy Participants: Carrot: Healthy adults with no history of difficulties with chewing or swallowing who were asked to chew and swallow a baby carrot.
- Healthy Participants: Cracker: Healthy adults with no history of chewing or swallowing difficulties who were asked to chew and swallow a single comfortable bite of a Carr's Table Water Cracker.
- Healthy Participants: Cracker With Barium Paste: Healthy adults with no history of chewing or swallowing difficulties who were asked to chew and swallow a single comfortable bite of a Carr's Table Water Cracker smeared with barium paste.
- Healthy Participants: Gummy Candy: Healthy adults with no history of chewing or swallowing difficulties who were asked to chew and swallow a round, dome-shaped gummy candy (Squish Vegan Red Rose).
- Healthy Participants: Minced and Moist Barium Stimulus: Healthy adults with no history of chewing or swallowing difficulties who were asked to chew and swallow a single bolus of a minced and moist consistency barium stimulus.
- Healthy Participants: Soft and Bite-sized Barium Stimulus: Healthy adults with no history of chewing or swallowing difficulties who were asked to chew and swallow a single bolus of a soft-and-bite-sized barium food stimulus.
Arm/Group | Healthy Participants: Carrot | Healthy Participants: Cracker | Healthy Participants: Cracker With Barium Paste | Healthy Participants: Gummy Candy | Healthy Participants: Minced and Moist Barium Stimulus | Healthy Participants: Soft and Bite-sized Barium Stimulus
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
number of chewing cycles | 22 (11) | 15 (6) | 15 (4) | 28 (13) | 6 (3) | 11 (4)

2. Primary Outcome: Total Chewing Duration Per Bolus
Description: Using surface electromyography (sEMG) of the masseter muscle, we will count the total duration of chewing activity for a single comfortable bite of each bolus type.
Time Frame: Baseline (single timepoint only)
Population: Data for 3 additional participants could not be analyzed due to poor EMG signal quality.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Healthy Participants: Carrot | Healthy Participants: Cracker | Healthy Participants: Cracker With Barium Paste | Healthy Participants: Gummy Candy | Healthy Participants: Minced and Moist Barium Stimulus | Healthy Participants: Soft and Bite-sized Barium Stimulus
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
seconds | 14.7 (5.4) | 13 (4.3) | 12.4 (2.7) | 25.1 (10.5) | 5.8 (2.6) | 9.9 (2.3)

ADVERSE EVENTS:
Time Frame: 48 hours following data collection
Description: Participants to contact the study team and report any health complaints experienced after data collection, such as gastrointestinal discomfort
Arm/Group | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants (N=18)
Digestive complaints (Gastrointestinal disorders) | 1 (1) — Complaints of abdominal discomfort and diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT05594173/Prot_SAP_000.pdf